CLINICAL TRIAL: NCT03652753
Title: Prevention of Cartilage Cell Death Following a Pilon Fracture With Intra-articular Injection of N-Acetylcysteine (Pilon NAC)
Brief Title: Pilon Fracture With Intra-articular Injection of N-Acetylcysteine (Pilon NAC)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kyle Schweser MD, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011492
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Pilon Fracture
MeSH Terms: interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine (NAC) (Experimental): Injection of N-acetylcysteine at the time of external fixation
  Interventions: Drug: N-acetylcysteine
- Saline (Placebo Comparator): Injection of saline at the time of external fixation
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: N-acetylcysteine — 4 mL of a 20% solution of NAC will be injected into the ankle of patients with pilon fractures at the time of their external fixator surgery
  Arms: N-acetylcysteine (NAC)
Drug: Saline — 4 mL of a 20% solution of saline will be injected into the ankle of patients with pilon fractures at the time of their external fixator surgery
  Arms: Saline

SUMMARY:
High energy intra-articular fractures of the distal tibia, or Pilon fracture, is a devastating injury with multiple short and long term complications. The incidence of these injuries is increasing as survival rates after motor vehicle collisions increase. The current standard of care for high energy pilon fractures is to place an external fixator at the time of injury and then provide definitive internal fixation when the soft tissue envelope allows, which is usually around 10-14 days. Arguably, the most debilitating long term complication after a high energy pilon fracture is the development of post-traumatic osteoarthritis (PTOA), which occurs in 50% or more of pilon fractures within the first 2 years of surgery. The development of osteoarthritis occurs even in the presence of adequate restoration of the tibial plafond. Part of this issue lies in the fact that ankle joint cartilage is the thinnest of any major articular joint and sustains a great deal of damage at the time of injury. This impaction and injury initiates a cascade of events that ultimately result in cartilage cell death, or chondrolysis. Chondrolysis occurs via necrosis or apoptosis. Apoptosis occurs via a caspase pathway, while necrosis of chondrocytes likely occurs secondary to overproduction of reactive oxidant species (ROS). Recent animal models have demonstrated several things: chondrocyte death is highest along fracture lines, and likely undergo necrosis as opposed to apoptosis. The reason that PTOA likely occurs in such a high percentage of pilon fractures is because of this chondrolysis, and if a method can be developed to decrease the rate of chrondrocyte necrosis, then the rate of PTOA could potentially improve and improve patient outcomes overall. A recent bovine model examined the injection of N-acetylcysteine (NAC) after an intra-articular knee fracture and its effect on the cartilage cell viability. Their study demonstrated that chondrocyte cell viability after an injection of NAC within four hours of injury decreased chondrolysis from roughly 60% to about 30% at 48hrs. The effect was greater the closer to injury the injection occurred, and was statistically significant for 2 weeks. This indicates that free radical scavengers can potentially improve cartilage cell viability and help prevent the development of PTOA. No studies have been published on humans regarding injection of NAC after a fracture. However, a recent article examined the injection of NAC into osteoarthritic knees and found that it was effective in lowering certain cartilage degradation markers and was comparable to hyaluronic acid for both pain and function. NAC has been proven safe for both intra-articular injections and systemic injections in humans. Our study will focus on the improvement of cartilage cell viability with an injection of NAC. Our hypothesis is that the NAC intra-articular injection will increase the percentage of viable cartilage cell after sustaining a pilon fracture, when compared to a placebo injection of saline.

The goal of this study is to examine the effects of an intra-articular injection of the amino acid NAC on cartilage cells after an intra-articular fracture of the ankle joint. The long-term clinical goal of this research is to reduce the incidence of post-traumatic osteoarthritis in the ankle joint after fracture.

ELIGIBILITY:
Inclusion Criteria:

* Closed high energy pilon fracture requiring a staged procedure

Exclusion Criteria:

* Younger than 18
* Open fracture
* Intra-articular injury not requiring a staged procedure
* Allergy to NAC
* Wounds preventing safe intra-articular injection
* Unwilling to participate in the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cartilage Cell Viability | At time of definitive surgery
  During the definitive surgery we will take a cartilage biopsy and analyze for cell viability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States